CLINICAL TRIAL: NCT02747940
Title: Neurologic Signatures of Chronic Pain Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-10-001BC2015-11-001AC002B
Record Dates: First submitted 2016-04-01; First posted 2016-04-22 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Chronic Pain; Chronic Migraine; Fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- patients with chronic migraine (Experimental): flunarizine for patients with chronic migraine
  Interventions: Drug: flunarizine and/or pregabalin
- patients with fibromyalgia (Experimental): pregabalin for patients with fibromyalgia
  Interventions: Drug: flunarizine and/or pregabalin
- patients with chronic migraine and fibromyalgia (Experimental): flunarizine and pregabalin for patients with chronic migraine and myalgia
  Interventions: Drug: flunarizine and/or pregabalin

INTERVENTIONS:
Drug: flunarizine and/or pregabalin

SUMMARY:
"Brain signatures" as objective measures of acute pain have been characterized with functional magnetic resonance image and machine learning technology. As compared to acute pain, chronic pain leads to greater socioeconomic burden. However, measures for chronic pain remain subjective and suboptimal, and the brain signatures for chronic pain are largely unknown. Chronic migraine and fibromyalgia are two prototypes primary chronic pain disorders with high disability and intractability with prevalence of around 2% for both diseases. These two chronic pain disorders have shared clinical presentations (abnormal pain sensitivity, mood and sleep disorders), pathophysiology (central sensitization) and medical treatment (anti-depressants), despite different body parts are involved (head vs. whole body). The present integrated project aims to characterize both common and disease-specific brain signatures of chronic pain by investigating these two chronic pain disorders. Our findings may shed some light on the key mechanisms of pain chronification, and may pave the way for the optimization of diagnosis and prognostication, as well as formulation of personalized medicine in chronic pain, so as to improve life quality of these patients and to reduce socioeconomic loss.

The present project includes three interdisciplinary sub-projects (plus one animal study, not listed here):

A: Clinical studies for chronic migraine and fibromyalgia: endophenotypes and pain chronification B: Functional neuroimaging of chronic pain: multimodal quantitative analysis of brain connectomes C. Data stream mining technology for multimodal physiological signals of chronic pain: real-time tracking and clinical correlation

The specific aims of the present projects include:

1. Identification of common and disease-specific brain signatures for chronic pain (sub-projects A, B, C)
2. Investigation of clinical indicators with predictive values by machine learning analysis of big data (sub-projects A, B, C)
3. Elucidation of the specific anatomical structures or neural networks underpinning pain chronification based on clinical neuroimaging (sub-projects A, B) In this 1st-year pilot study of the 4-year longitudinal study, we will establish experimental platforms for each sub-project, start to recruit participants and perform endophenotyping, as well as have a preliminary integration for sub-projects A, B and C.

ELIGIBILITY:
Inclusion Criteria:

* Control: devoid of any systemic or neurological diseases
* Chronic migraine: by ICHD-III (International Classification of Headache Disorder) criteria
* Fibromyalgia: by ACR (American College of Rheumatology) 2010 criteria

Exclusion Criteria:

* history of major systemic illness, including uncontrolled hypertension, diabetes, chronic renal insufficiency, autoimmune diseases or malignancies
* history of neurological disorders which might affect sensation such as previous stroke or peripheral neuropathy
* history of substance abuse (except painkillers)
* heavy smokers (with a daily consumption >20 cigarettes)
* pregnancy or lactation
* any contraindication for magnetic resonance imaging (MRI)
* and any obvious infection or inflammation over a period of at least 1 month before the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
clinical improvement after treatment (1) headache/pain intensity [NRS, numeric rating scale] | 4 months
  clinical improvement (headache/pain intensity) after treatment unit: NRS (numeric rating scale, 0-10) analysis: comparing the mean headache/pain intensity in each month after treatment (M1/M2/M3/M4) to that before treatment (M-1)
clinical improvement after treatment (2) headache/pain frequency [attacks per month] | 4 months
  clinical improvement (headache/pain frequency) after treatment unit: attacks per month analysis: comparing the mean headache/pain frequency in each month after treatment (M1/M2/M3/M4) to that before treatment (M-1)
clinical improvement after treatment (3) headache/pain duration [hours per day] | 4 months
  clinical improvement (headache/pain duration) after treatment unit: hours/day analysis: comparing the mean headache/pain duration (hours/day) in each month after treatment (M1/M2/M3/M4) to that before treatment (M-1)

SECONDARY OUTCOMES:
EEG change after treatment | 4 months
  Linear and nonlinear analysis of EEG before and after treatment
  * Three EEG session will be arranged. The first one is done before treatment, and the 2nd/3rd one will be done after a 2-month/4-month treatment course, respectively.
  * The EEG analyses include linear (eg: power spectrum, coherence, functional connectivity) analyses as well as non-linear (eg: entropy) analyses.
sensory and pain threshold change after treatment | 2 months
  Using quantitative sensory testing (QST) to evaluate the sensory and pain threshold before and after treatment
  * Three QST session will be arranged. The first one is done before treatment, and the 2nd/3rd one will be done after a 2-month/4-month treatment course, respectively.
  * Equipment: electric von Fray filaments
  * unit: gram
Autonomic function change after treatment | 2 months
  Using heart rate variability (HRV) to evaluate autonomic function before and after treatment
  * Three HRV session will be arranged. The first one is done before treatment, and the 2nd/3rd one will be done after a 2-month/4-month treatment course, respectively.
  * The HRV analyses include time-domain (eg: mean heart rate and its variation, mean R-R interval and its variation), and also frequency domain analysis (eg: power spectrum)

CONTACTS AND LOCATIONS:
Overall Officials: Shuu-Jiun Wang, M.D., Principal Investigator — Neurological Institute, Taipei Veterans General Hospital
Locations (1):
- Headache Center, Teipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuang CH, Li JY, King JT, Chen WT, Chen SP, Wang YF, Liu HY, Hsiao FJ, Pan LH, Wang SJ, Lai KL. Abnormal heart rate variability and its application in predicting treatment efficacy in patients with chronic migraine: An exploratory study. Cephalalgia. 2023 Oct;43(10):3331024231206781. doi: 10.1177/03331024231206781. PMID 37851663
- [Derived] Pan LH, Chen WT, Wang YF, Chen SP, Lai KL, Liu HY, Hsiao FJ, Wang SJ. Resting-state occipital alpha power is associated with treatment outcome in patients with chronic migraine. Pain. 2022 Jul 1;163(7):1324-1334. doi: 10.1097/j.pain.0000000000002516. Epub 2021 Oct 13. PMID 35708466
- [Derived] Pan LH, Wang YF, Ling YH, Lai KL, Chen SP, Chen WT, Treede RD, Wang SJ. Pain sensitivities predict prophylactic treatment outcomes of flunarizine in chronic migraine patients: A prospective study. Cephalalgia. 2022 Aug;42(9):899-909. doi: 10.1177/03331024221080572. Epub 2022 Apr 11. PMID 35400174
- [Derived] Hsiao FJ, Chen WT, Liu HY, Wang YF, Chen SP, Lai KL, Hope Pan LL, Coppola G, Wang SJ. Migraine chronification is associated with beta-band connectivity within the pain-related cortical regions: a magnetoencephalographic study. Pain. 2021 Oct 1;162(10):2590-2598. doi: 10.1097/j.pain.0000000000002255. PMID 34534180
- [Derived] Hsiao FJ, Chen WT, Ko YC, Liu HY, Wang YF, Chen SP, Lai KL, Lin HY, Coppola G, Wang SJ. Neuromagnetic Amygdala Response to Pain-Related Fear as a Brain Signature of Fibromyalgia. Pain Ther. 2020 Dec;9(2):765-781. doi: 10.1007/s40122-020-00206-z. Epub 2020 Oct 22. PMID 33090368